CLINICAL TRIAL: NCT01941693
Title: Novel Treatments for Alcohol Dependence: A Randomized Controlled Trial of Structured Stepped-care Intervention for Psychiatric Comorbidity
Brief Title: A Randomized Controlled Trial of Structured Stepped-care Intervention for Psychiatric Comorbidity
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: South West Sydney Local Health District (Other)
Collaborators: University of Sydney (Other)
Responsible Party: Principal Investigator, Professor Paul Haber, Medical Director, South West Sydney Local Health District
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: X05-0279
Record Dates: First submitted 2013-09-05; First posted 2013-09-13 (Estimated); Last update posted 2013-09-13 (Estimated); Status verified 2013-09

CONDITIONS: Alcohol Dependence; Anxiety; Depression
Keywords: alcohol; anxiety; depression; comorbidity; CBT
MeSH Terms: conditions — Alcoholism; Anxiety Disorders; Depression | interventions — Delivery of Health Care, Integrated

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Integrated care (Experimental): Integrated care:
  Intervention for co-morbid alcohol dependence and anxiety or mood disorder. Trained therapists will deliver specific Cognitive Behavioural Therapy based upon interventions that have been supported by randomised controlled trials for alcohol use, anxiety, and depressive disorders.
  Interventions: Behavioral: Integrated care
- Usual care (Active Comparator): Usual care
  Interventions: Behavioral: Usual care

INTERVENTIONS:
Behavioral: Integrated care — Intervention for co-morbid alcohol dependence and anxiety or mood disorder. Trained therapists will deliver specific Cognitive Behavioural Therapy based upon interventions that have been supported by randomised controlled trials for alcohol use, anxiety, and depressive disorders.
  Arms: Integrated care
Behavioral: Usual care — Counselling for all subjects will continue in accord with standard practice. Currently, programs of brief individualized motivation enhancement therapy (feedback of assessment findings, reinforcement, empathy, client's own motivation) are available.
  Arms: Usual care

SUMMARY:
There is a high rate of psychological comorbidity in people suffering from alcohol dependence. There is a need for an effective integrated treatment for alcohol dependence and comorbid anxiety or depression. This study will test the efficacy of a novel integrated intervention for comorbid alcohol dependence and anxiety or mood disorder.

DETAILED DESCRIPTION:
In summary, the specific aims of this project are:

1. To assess the effectiveness of a novel stepped care intervention for alcohol dependent patients with co-morbid anxiety and/or depression compared to usual treatment for alcohol dependence in promoting abstinence from alcohol and increased quality of life and in reducing symptoms of anxiety and depression.
2. To describe important factors relating to the maintenance of alcohol-related psychiatric comorbidity.

Step 1: All subjects will complete 12 weeks of pharmacotherapy (n = 120) on naltexone (50 mg, 1 tablet daily), acamprosate (333 mg, 2 tablets 3 times daily, reduced to 4/day for women <65kg), or a combination of the two. After a 3 week stabilization period, subjects will undergo complete formal assessment for anxiety and depression. Those subjects with a diagnosis of anxiety or depressive disorder regardless of drinking outcome will be offered the next step of care and followed up at 12-16 weeks.

Step 2: Subjects to undergo the next step of care (n = 30 per group, 60 in total) will be randomized by referring to the consecutively assigned subject identification number to a matched numbered envelope containing a random assignment card. Randomization will be stratified according to concomitant SSRI use. The treatment groups will be:

1. Intervention for comorbid anxiety or depression, and
2. Usual counseling care.

ELIGIBILITY:
Inclusion Criteria for Step 1:

* alcohol dependence according to DSM-IV criteria, with alcohol as the subject's drug of choice,
* age 18-65,
* adequate cognition and English language skills to give valid consent and complete research interviews (as assessed by the mini mental state examination),
* willingness to give written consent,
* abstinence from alcohol for between 3 and 21 days (standard clinical criteria for use of acamprosate or naltrexone),
* resolution of any clinically evident alcohol withdrawal (score 0-1 on RPA hospital alcohol withdrawal scale), and a positive score on the initial comorbidity suspicion checklist (CSC).

Exclusion Criteria for Step 1:

* sensitivity to study medications or therapy with these drugs within 6 months,
* active major psychiatric disorder associated with significant suicide risk,
* pregnancy or lactation,
* advanced liver disease (hepatocellular failure, variceal bleeding, ascites or encephalopathy),
* other serious medical illness that would interfere with adherence to the study protocol.

Entry criteria to step 2:

* Completion of 3 weeks on acamprosate and/or natlrexone and/or, resolution of any clinically evident alcohol withdrawal (score 0-1 on RPA hospital alcohol withdrawal scale),
* case formulation and diagnosis for anxiety or depression (see below).

Exclusion criteria 2:

* Non-compliance on acamprosate and/or naltrexone,
* alcohol consumption at baseline levels,
* resolution of clinically evident anxiety or depression as assessed by the case formulation (see below). These patients will be offered further treatment

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 86 (Actual)
Dates: Start 2007-03; Primary Completion 2010-12 (Actual); Study Completion 2013-03 (Actual)

PRIMARY OUTCOMES:
Alcohol consumption | 12 weeks
  Time to relapse (>5 drinks on any one day)
Time to lapse | 12 weeks
  time to consumption of any alcohol (lapse) identified by self-reported alcohol consumption
amount of alcohol consumption | 12 weeks
  expressed as the average consumption per drinking day

SECONDARY OUTCOMES:
Improvement in depressive or anxiety symptoms | 12 weeks
  DASS 21
Diagnosis severity | 16 weeks
  clinician rated severity from ADIS-IV and HDRS on anxiety and depressive diagnoses.

CONTACTS AND LOCATIONS:
Overall Officials: Andrew Baillie, Principal Investigator — Macquarie University; Paul Haber, Principal Investigator — University of Sydney
Locations (1):
- Drug Health Services, Royal Prince Alfred Hospital, Sydney, New South Wales, Australia

REFERENCES:
- [Derived] Morley KC, Baillie A, Leung S, Sannibale C, Teesson M, Haber PS. Is Specialized Integrated Treatment for Comorbid Anxiety, Depression and Alcohol Dependence Better than Treatment as Usual in a Public Hospital Setting? Alcohol Alcohol. 2016 Jul;51(4):402-9. doi: 10.1093/alcalc/agv131. Epub 2015 Dec 15. PMID 26672793
- [Derived] Morley KC, Baillie A, Sannibale C, Teesson M, Haber PS. Integrated care for comorbid alcohol dependence and anxiety and/or depressive disorder: study protocol for an assessor-blind, randomized controlled trial. Addict Sci Clin Pract. 2013 Nov 19;8(1):19. doi: 10.1186/1940-0640-8-19. PMID 24245491